CLINICAL TRIAL: NCT04323787
Title: Viral Infection and Respiratory Illness Universal Study[VIRUS]: COVID-19 Registry and Validation of C2D2 (Critical Care Data Dictionary)
Brief Title: Viral Infection and Respiratory Illness Universal Study[VIRUS]: COVID-19 Registry
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Society of Critical Care Medicine (Other); Boston University (Other)
Responsible Party: Principal Investigator, Juan Pablo Domecq Garces, Principal Investigator, Mayo Clinic
Other Study IDs: 20-002610
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Coronavirus
Keywords: COVID19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COVID19 test positive/pending or high clinical suspicion: COVID19 test positive/pending/high clinical suspicion- patient admitted to hospital
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — No Intervention
  Other Names: No Intervention

SUMMARY:
Researchers are creating a real time COVID-19 registry of current ICU/hospital care patterns to allow evaluations of safety and observational effectiveness of COVID-19 practices and to determine the variations in practice across hospitals.

DETAILED DESCRIPTION:
Investigators aim is to create a real time COVID-19 registry of current ICU/hospital care patterns to allow evaluations of safety and observational effectiveness of COVID-19 practices and to determine the variations in practice across hospitals.

Such a set of standards would increase the quality of single and multi-center studies, national registries as well as aggregation syntheses such as meta-analyses. It will also be of utmost importance in tiring times of public health emergencies and will help understand practice variability and outcomes during COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 PCR positive (within 7 days)
* COVID-19 PCR pending
* COVID-19 high clinical suspicion

Exclusion Criteria:

* Patient without Prior Research Authorization (applicable to Mayo Clinic sites)
* Non COVID-19 related admissions
* Repeated Admission to ICUs/Hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COVID-19 Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
ICU and hospital mortality of COVID-19 patients | 7 days
  Primary outcome will be to measure ICU and hospital mortality up to 7 days of COVID-19 patients

SECONDARY OUTCOMES:
30 days mortality | 30 days
  Secondary outcome will be to measure 30 days mortality from Hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pablo Domecq Garces, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Society of Critical Care Medicine (150+ sites), Chicago, Illinois
  - Rahul Kashyap, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Truwit JD, Fleming K, Nanchal RS. Empowering Respiratory Therapists to Restrict Nebulized 3% Saline and N-Acetylcysteine During Mechanical Ventilation. Respir Care. 2025 Aug;70(8):937-945. doi: 10.1089/respcare.12586. Epub 2025 Feb 24. PMID 40028879
- [Derived] Tekin A, Qamar S, Sharma M, Singh R, Malinchoc M, Bansal V, Deo N, Bogojevic M, Valencia-Morales DJ, Zec S, Zorko-Garbajs N, Sharma N, Lal A, Sanghavi DK, Cartin-Ceba R, Khan SA, La Nou AT, Cherian A, Zabolotskikh IB, Kumar VK, Kashyap R, Walkey AJ, Domecq JP, Yadav H, Gajic O, Odeyemi YE; Society of Critical Care Medicine Discovery Viral Infection and Respiratory Illness Universal Study (VIRUS): COVID-19 Registry Investigator Group. Development and Validation of an Acute Respiratory Distress Syndrome Prediction Model in Coronavirus Disease 2019: Updated Lung Injury Prediction Score. Mayo Clin Proc. 2023 May;98(5):736-747. doi: 10.1016/j.mayocp.2022.11.021. Epub 2022 Dec 30. PMID 37028977
- [Derived] Gupta N, Settle L, Brown BR, Armaignac DL, Baram M, Perkins NE, Kaufman M, Melamed RR, Christie AB, Danesh VC, Denson JL, Cheruku SR, Boman K, Bansal V, Kumar VK, Walkey AJ, Domecq JP, Kashyap R, Aston CE; Society of Critical Care Medicine Discovery Viral Infection and Respiratory Illness Universal Study (VIRUS): COVID-19 Registry Investigator Group. Association of Renin Angiotensin Aldosterone System Inhibitors and Outcomes of Hospitalized Patients With COVID-19. Crit Care Med. 2022 Oct 1;50(10):e744-e758. doi: 10.1097/CCM.0000000000005627. Epub 2022 Jul 27. PMID 35894609
- [Derived] Garcia MA, Johnson SW, Sisson EK, Sheldrick CR, Kumar VK, Boman K, Bolesta S, Bansal V, Bogojevic M, Domecq JP, Lal A, Heavner S, Cheruku SR, Lee D, Anderson HL, Denson JL, Gajic O, Kashyap R, Walkey AJ; from the Society of Critical Care Medicine's Discovery Viral Infection and Respiratory Illness Universal Study Investigators. Variation in Use of High-Flow Nasal Cannula and Noninvasive Ventilation Among Patients With COVID-19. Respir Care. 2022 Aug;67(8):929-938. doi: 10.4187/respcare.09672. Epub 2022 Jun 7. PMID 35672139
- [Derived] Sayed IA, Bhalala U, Strom L, Tripathi S, Kim JS, Michaud K, Chiotos K, Dapul HR, Gharpure VP, Bjornstad EC, Heneghan JA, Irby K, Montgomery V, Gupta N, Gupta M, Boman K, Bansal V, Kashyap R, Walkey AJ, Kumar VK, Gist KM; VIRUS Investigators. Gastrointestinal Manifestations in Hospitalized Children With Acute SARS-CoV-2 Infection and Multisystem Inflammatory Condition: An Analysis of the VIRUS COVID-19 Registry. Pediatr Infect Dis J. 2022 Sep 1;41(9):751-758. doi: 10.1097/INF.0000000000003589. Epub 2022 May 27. PMID 35622434
- [Derived] Turek JR, Bansal V, Tekin A, Singh S, Deo N, Sharma M, Bogojevic M, Qamar S, Singh R, Kumar V, Kashyap R. Lessons From a Rapid Project Management Exercise in the Time of Pandemic: Methodology for a Global COVID-19 VIRUS Registry Database. JMIR Res Protoc. 2022 Mar 15;11(3):e27921. doi: 10.2196/27921. PMID 34762062
- [Derived] Kirkup C, Pawlowski C, Puranik A, Conrad I, O'Horo JC, Gomaa D, Banner-Goodspeed VM, Mosier JM, Zabolotskikh IB, Daugherty SK, Bernstein MA, Zaren HA, Bansal V, Pickering B, Badley AD, Kashyap R, Venkatakrishnan AJ, Soundararajan V. Healthcare disparities among anticoagulation therapies for severe COVID-19 patients in the multi-site VIRUS registry. J Med Virol. 2021 Jul;93(7):4303-4318. doi: 10.1002/jmv.26918. Epub 2021 Mar 30. PMID 33666246
- [Derived] Domecq JP, Lal A, Sheldrick CR, Kumar VK, Boman K, Bolesta S, Bansal V, Harhay MO, Garcia MA, Kaufman M, Danesh V, Cheruku S, Banner-Goodspeed VM, Anderson HL 3rd, Milligan PS, Denson JL, St Hill CA, Dodd KW, Martin GS, Gajic O, Walkey AJ, Kashyap R. Outcomes of Patients With Coronavirus Disease 2019 Receiving Organ Support Therapies: The International Viral Infection and Respiratory Illness Universal Study Registry. Crit Care Med. 2021 Mar 1;49(3):437-448. doi: 10.1097/CCM.0000000000004879. PMID 33555777
- See also: SCCM Discovery VIRUS COVID19 Information Webpage — https://www.sccm.org/VIRUS